CLINICAL TRIAL: NCT05036889
Title: A 16-week Randomized Evaluation of the Impact of Mind.Px Application on Response to Biologic Treatment in Patients Suffering From Plaque Psoriasis Through Clinical Utility and Health Outcomes.
Acronym: MATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mindera Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MND-21-MKPs-02
Record Dates: First submitted 2021-08-17; First posted 2021-09-08 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MND (Experimental): Subject's physician in this group will be using the Mind.Px report as a treatment reference for prescribing the subject's biologic.
  Interventions: Diagnostic Test: Mind.Px Report
- TAU (No Intervention): Treatment as usual. This group will have the biologic prescribed with results given to the physician at the end of the subject's participation and will not be used as a reference for the subject's treatment.

INTERVENTIONS:
Diagnostic Test: Mind.Px Report — Use of Mind.Px report as a reference for potential better matching of biologics to patients.
  Arms: MND

SUMMARY:
This protocol describes randomized, multicenter, blinded (subjects), 16-week, controlled study in parallel balanced groups of psoriasis (Ps) patients to evaluate the impact of Mind.Px on response to biologic treatments. Patients enrolled in this study will be required to have diagnosis of Ps and a total score ≥10 on the PASI and the identified study-lesion must have a PGA severity ≥3 on a 5-point scale of 0 to 4.

Patients suffering from Ps will be enrolled in the study and randomized on a 1:1 basis to treatment as usual (TAU) or to treatment decision utilizing Mind.Px (MND). Both groups will have a dermal patch applied and analyzed. The TAU group will not be provided the results of the dermal patch until the end of the last study visit. The MND group will be provided the results of the dermal patch upon the completion of the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have the ability to understand and sign written informed consent.
2. Subject must be an adult male or female adult who is ≥ 18 years of age at the time of screening.
3. Subject must be diagnosed with plaque psoriasis by either a dermatologist or a rheumatologist, with the affected area of ≥ 2 centimeters in diameter (study-lesion).
4. Subjects must be treated with an anti-IL-17, anti-IL-23, or an anti TNF-α biologic
5. Subject must abstain from the use of any treatment to the identified study-lesion after screening until the baseline visit (this includes biologic treatments until after the dermal patch sample has been collected).
6. Subjects must abstain from the use of steroid or any topical treatment to the identified study lesion from screening till the last study visit.
7. Subjects must have a baseline PASI ≥10 and the identified study-lesion must have a PGA severity ≥3 on a 5-point scale of 0 to 4.
8. Agree to abide by the study protocol and its restrictions and be able to complete all aspects of the study, including all visits and tests.

Exclusion Criteria:

1. Subject is unable or unwilling to give written informed consent and/or to comply with study procedures.
2. Subject has had new usage of topical psoriasis treatments within 2 weeks prior to screening study visit (these concomitant immunomodulatory treatments such as corticosteroid/calcineurin inhibitors).
3. Subjects currently treated with Hydroxychloroquine (Plaquenil).
4. Subjects has had usage of anti TNF-α, IL-12/23, IL-17, IL-23, JAK inhibitor, or T-cell activation inhibitor, therapy within 2 weeks prior to baseline, unless otherwise approved by Sponsor.
5. More than 2 prior treatments with a biologic therapy.
6. Subjects with a BMI ≥40 and a diagnosis of Class III (Severe) Obesity (or solely a diagnosis of Class III (Severe) Obesity).
7. Any change in biologic medication (including change in dosage) between screening and randomization.
8. No phototherapy or other oral systemic therapy (acitretin, ciclosporin, methotrexate, apremilast, fumarate, oral JAK inhibitor, or T-cell activation inhibitor) at least 2 weeks before baseline and throughout study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-24 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of Mind.Px on response to biologic treatment as judged by the mean change in the Psoriasis Area Severity index (PASI) score from baseline to end of Week 16 of the study. | 16 weeks
  Evaluate the impact of Mind.Px on response to biologic treatment as judged by the mean change in the Psoriasis Area Severity index (PASI) score from baseline to end of Week 16 of the study.

SECONDARY OUTCOMES:
Mean change in the Physician Global Assessment (PGA) by the Body Surface Area (BSA), or Dermatology Life Quality Index (DLQI) from baseline to end of Week 16 of the study | 16 weeks
  Mean change in the Physician Global Assessment (PGA) by the Body Surface Area (BSA), or Dermatology Life Quality Index (DLQI) from baseline to end of Week 16 of the study

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strober BE, Bukhalo M, Armstrong AW, Pariser D, Kircik L, Johnson B, Montgomery P 3rd, Dickerson TJ. Clinical Utility Findings of a Transcriptomic Psoriasis Biologic Test Demonstrate Altered Physician Prescribing Behavior and Improved Patient Outcomes. Dermatol Ther (Heidelb). 2025 Jul;15(7):1787-1796. doi: 10.1007/s13555-025-01441-y. Epub 2025 May 11. PMID 40349264